CLINICAL TRIAL: NCT00887159
Title: A Randomized Phase II Study of Cisplatin and Etoposide in Combination With Either Hedgehog Inhibitor GDC-0449 or IGF-1R MOAB IMC-A12 for Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: A Randomized Phase II Study of Cisplatin and Etoposide in Combination With Either Hedgehog Inhibitor GDC-0449 or IGF-1R MOAB IMC-A12 for Patients With Extensive Stage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01917; NCI-2011-01917 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 09-0679; ECOG-E1508; CDR0000640898; E1508 (Other: ECOG-ACRIN Cancer Research Group); E1508 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2015-07-29 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Extensive Stage Small Cell Lung Carcinoma; Recurrent Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; cixutumumab; Etoposide; HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (CE) (Active Comparator): Patients receive cisplatin IV over 1-2 hours on day 1 and etoposide IV over 1-2 hours on days 1-3. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Etoposide; Other: Laboratory Biomarker Analysis
- Arm B (CE + GDC-0449) (Experimental): Patients receive cisplatin and etoposide as in Arm A and vismodegib PO QD on days 1-21. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive vismodegib alone QD in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Vismodegib
- Arm C (CE + IMC-A12) (Experimental): Patients receive cisplatin and etoposide as in Arm A and cixutumumab IV over 1 hour on days 1, 8, and 15. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive cixutumumab alone once weekly in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Biological: Cixutumumab; Drug: Etoposide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Biological: Cixutumumab — Given IV
  Other Names: Anti-IGF-1R Recombinant Monoclonal Antibody IMC-A12; IMC-A12
  Arms: Arm C (CE + IMC-A12)
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC-0449; Hedgehog Antagonist GDC-0449
  Arms: Arm B (CE + GDC-0449)

SUMMARY:
This randomized phase II trial studies cisplatin and etoposide to see how well they work when given with or without Hedgehog inhibitor GDC-0449 (vismodegib) or IGF-1R MOAB IMC-A12 (cixutumumab) in treating patients with extensive-stage small cell lung cancer. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Etoposide may slow the growth of tumor cells by blocking some of the enzymes needed for cell growth. Vismodegib may slow the growth of tumor cells. Monoclonal antibodies, such as cixutumumab, may interfere with the ability of tumor cells to grow and spread. It is not yet known whether giving cisplatin and etoposide are more effective when given together with vismodegib or cixutumumab in treating small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the progression-free survival (PFS) of patients with extensive stage small cell lung cancer (SCLC-ED) treated with cisplatin and etoposide (CE), CE with hedgehog (HH) inhibitor GDC-0449 (vismodegib), and CE with insulin-like growth factor-1 receptor (IGF-1R) monoclonal antibody (IMC-A12) (cixutumumab).

SECONDARY OBJECTIVES:

I. To evaluate response rate, overall survival, and toxicity for each arm. II. To explore putative correlates of clinical benefit from combination therapy in tumor and circulating tumor cells in patients treated on this protocol.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM A (CE): Patients receive cisplatin (75 mg/m^2) intravenously (IV) over 1-2 hours on day 1 and etoposide (100 mg/m^2) IV over 1-2 hours on days 1-3. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

ARM B (CE +GDC-0449): Patients receive cisplatin and etoposide as in Arm A and vismodegib (GDC-0449; 150 mg tablet) orally (PO) once daily (QD) on days 1-21. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive vismodegib alone QD in the absence of disease progression or unacceptable toxicity.

ARM C (CE + IMC-A12): Patients receive cisplatin and etoposide as in Arm A and cixutumumab (IMC-A12; 6 mg/kg) IV over 1 hour on days 1, 8, and 15. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive cixutumumab alone once weekly in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small cell lung cancer (SCLC)
* Extensive stage SCLC

  * Extensive stage disease: the extensive disease classification for this protocol includes all patients with disease sites not defined as limited stage; limited stage disease category includes patients with disease restricted to one hemithorax with regional lymph node metastases, including hilar, ipsilateral and contralateral mediastinal, and/or ipsilateral supraclavicular nodes; extensive disease patients are defined as those patients with extrathoracic metastatic disease, malignant pleural effusion, bilateral or contralateral supraclavicular adenopathy
* Measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST); baseline measurements and evaluations of all sites of disease must be obtained =< 4 weeks prior to randomization
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase)/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase) =< 3 x institutional ULN (=< 5 x ULN if liver function test [LFT] elevations are due to liver metastases)
* Creatinine =< 1.5 x institutional ULN OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels > 1.5 x institutional ULN
* Leukocytes >= 3,000/mm^3
* Hemoglobin >= 9 g/dL
* Fasting serum glucose < 120 mg/dL or below institutional ULN =< 7 days prior to protocol randomization
* Patients with central nervous system (CNS) metastases will be eligible if they have completed a course of CNS radiotherapy and have stable neurologic function for a minimum of 28 days prior to study randomization; radiotherapy must have been completed a minimum of 28 days prior to randomization, and patients must have recovered from any adverse events related to the radiotherapy (except alopecia and grade 1 neuropathy) and have stable neurologic function for a minimum of 28 days prior to study randomization

  * NOTE: the use of prophylactic cranial irradiation (recommended dose 25 Gy) in those who completed protocol chemotherapy and have a response (in the absence of progressive disease [PD]) is allowed; for patients on Arms B and C, GDC-0449 and IMC-A12 will be held while patient is receiving prophylactic cranial irradiation (PCI); these agents can be reinstituted after PCI is completed
* Women of child-bearing potential (WCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation

  * WCBP must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse; the two methods of reliable contraception must include one highly effective method (i.e., intrauterine device [IUD], hormonal [birth control pills, injections, or implants], tubal ligation, partner?s vasectomy) and one additional effective (barrier) method (i.e., latex condom, diaphragm, cervical cap); WCBP must be referred to a qualified provider of contraceptive methods if needed

    * NOTE: the WCBP randomized to Arm B must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following two additional time periods related to this study: 1) while participating in the study; and 2) for at least 12 months after discontinuation from the study
  * Before starting the study drugs, all WCBP must have a negative pregnancy test (sensitivity of at least 50 mIU/mL); the pregnancy test must be performed within 10-14 days prior to randomization

    * NOTE: the WCBP randomized to Arm B must have a second pregnancy test performed within the 24 hours prior to the start of the GDC-0449; the subject may not receive GDC-0449 until the investigator has verified that the results of these pregnancy tests are negative
  * The WCBP randomized to Arm B will be warned that sharing the study drug is prohibited and will be counseled about pregnancy precautions and potential risks or fetal exposure; she must also agree to abstain from donating blood during study participation and at least 12 months after discontinuation from the study drug

    * NOTE: male subjects randomized to Arm B must agree to use a latex condom during sexual contact with WCBP while participating in the study and for at least 12 months following discontinuation from the study even if he has undergone a successful vasectomy
  * Male subjects randomized to Arm B will be warned that sharing study drug is prohibited and will be counseled about pregnancy precautions and potential risks of fetal exposure; male subjects must agree to abstain from donating blood, semen, or sperm during study participation and for at least 3 months after discontinuation from the study drug

Exclusion Criteria:

* Pregnant or breastfeeding; all WCBP must have a blood test within 10-14 days prior to randomization to rule out pregnancy
* Prior chemotherapy or biologic therapy for SCLC; patients with prior radiation may be eligible or after palliative radiotherapy for other sites of disease; patients receiving prior radiation cannot start therapy within 14 days after completion of radiation, and must have recovered from adverse events attributed to radiation; no previous irradiation to the only site of measurable or evaluable disease, unless that site had subsequent evidence of progression
* Receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biological composition to GDC-0449 and IMC-A12 or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy
* Poorly controlled diabetes mellitus; patients with a history of diabetes mellitus are allowed to participate, provided that their blood glucose is within normal range (fasting < 120 mg/dL or below institutional upper limit of normal) and that they are on a stable dietary or therapeutic regimen for this condition
* Patients with major surgery, hormonal therapy (other than replacement), within 4 weeks prior to entering the study or those who have not recovered from adverse events
* Prior treatment with other agents targeting the IGFR or the Hedgehog signaling pathway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2009-07-16 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Belani, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (301):
- United States (301):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Presence Saint Joseph Hospital-Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - The Memorial Hospital at Easton, Easton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - New York Oncology Hematology PC - Albany, Albany, New York
  - New York Oncology Hematology PC -Albany Medical Center, Albany, New York
  - New York Oncology Hematology PC - Amsterdam, Amsterdam, New York
  - New York Oncology Hematology PC - Clifton Park, Clifton Park, New York
  - New York Oncology Hematology PC-Hudson, Hudson, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - New York Oncology Hematology PC - Rexford, Rexford, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Oncology Hematology PC - Troy, Troy, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - West Virginia University Charleston, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Columbia Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- See also: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG member institutions between July, 16, 2009 and August 12, 2011.
Groups:
- Arm A (CE): Patients receive cisplatin (75 mg/m2) intravenously (IV) over 1-2 hours on day 1 and etoposide (100 mg/m2) IV over 1-2 hours on days 1-3. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  cisplatin: Given IV
  etoposide: Given IV
- Arm B (CE+GDC-0449): Patients receive cisplatin and etoposide as in Arm A and vismodegib (GDC-0449; 150 mg tablet) orally (PO) once daily (QD) on days 1-21. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive vismodegib alone QD in the absence of disease progression or unacceptable toxicity.
  vismodegib: Given PO
  cisplatin: Given IV
  etoposide: Given IV
- Arm C (CE+IMC-A12): Patients receive cisplatin and etoposide as in Arm A and cixutumumab (IMC-A12; 6 mg/kg) IV over 1 hour on days 1, 8, and 15. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive cixutumumab alone once weekly in the absence of disease progression or unacceptable toxicity.
  cixutumumab: Given IV
  cisplatin: Given IV
  etoposide: Given IV
Period: Overall Study
Arm/Group | Arm A (CE) | Arm B (CE+GDC-0449) | Arm C (CE+IMC-A12)
Started | 56 | 56 | 56
Patients Who Started Assigned Treatment | 53 | 53 | 52
Eligible and Treated Patients | 48 | 52 | 52
Eligible/Treated Pts With CTCs Results | 40 | 42 | 38
Completed | 27 | 0 (Treatment continued until disease progression or unacceptable toxicity.) | 0 (Treatment continued until disease progression or unacceptable toxicity.)
Not Completed | 29 | 56 | 56
Not completed — Disease progression | 6 | 39 | 33
Not completed — Adverse Event | 3 | 4 | 17
Not completed — Death | 2 | 2 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 2
Not completed — Alternative therapy | 2 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Sympomatic deterioration | 1 | 0 | 0
Not completed — Treatment delayed | 1 | 1 | 0
Not completed — Pt had PD but was SD when re-measured | 0 | 1 | 0
Not completed — Received more tx instead of observation | 1 | 0 | 0
Not completed — Ineligible | 5 | 1 | 0
Not completed — Never started assigned therapy | 3 | 3 | 4

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (CE) | Arm B (CE+GDC-0449) | Arm C (CE+IMC-A12) | Total
Number analyzed (Participants) | 48 | 52 | 52 | 152
Age, Continuous [Median (Full Range); unit: years] | 61 [38 to 77] | 64 [52 to 87] | 64 [45 to 83] | 63 [38 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 25 | 76
  Male | 23 | 26 | 27 | 76
Region of Enrollment [Number; unit: participants]
  United States | 48 | 52 | 52 | 152

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from randomization to death or disease progression, whichever occurred first. Patients who were alive at the time of analysis are censored at the date at which they are last known to be alive and progression-free.
Time Frame: Assessed every 6 weeks while on treatment or observation; follow-up after discontinuation of treatment or observation: every 3 months if patient is < 2 years from study entry, every 6 months if patient is 2-3 years from study entry
Population: Eligible and treated patients.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm A (CE): Patients receive cisplatin (75 mg/m2) intravenously (IV) over 1-2 hours on day 1 and etoposide (100 mg/m2) IV over 1-2 hours on days 1-3. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
- Arm B (CE+GDC-0449): Patients receive cisplatin and etoposide as in Arm A and vismodegib (GDC-0449; 150 mg tablet) orally (PO) once daily (QD) on days 1-21. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive vismodegib alone QD in the absence of disease progression or unacceptable toxicity.
- Arm C (CE+IMC-A12): Patients receive cisplatin and etoposide as in Arm A and cixutumumab (IMC-A12; 6 mg/kg) IV over 1 hour on days 1, 8, and 15. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive cixutumumab alone once weekly in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A (CE) | Arm B (CE+GDC-0449) | Arm C (CE+IMC-A12)
Number analyzed (Participants) | 48 | 52 | 52
months | 4.4 [3.6 to 5.5] | 4.4 [4.1 to 5.4] | 4.6 [4.4 to 5.5]
Statistical Analysis 1: Comparison: Arm A (CE) vs Arm B (CE+GDC-0449); There are 2 primary comparisons and each involves comparing the experimental arms (B, C) to the control arm (A). Accrual goal was 54 patients per arm. With a 1-sided 0.1 level logrank test for each test, we have 90% power to detect a 42% reduction in the PFS hazard rate of 0.139 to 0.082 (corresponding to an improvement in median PFS of 5 months to 8.5 months) with 18-month accrual and 12-month follow-up; assuming exponential survival. For each test, 94 events are needed to achieve this power; Test type: Superiority or Other; p = 0.45, Regression, Cox — P-value is one-sided; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.65 to 1.47] — The hazard ratio was derived comparing Arm B to Arm A
Statistical Analysis 2: Comparison: Arm A (CE) vs Arm C (CE+IMC-A12); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.48, Regression, Cox — P-value is one-sided; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.66 to 1.48] — Hazard ratio was derived comparing Arm C to Arm A

2. Secondary Outcome: Response Rate
Description: Response rate is defined as number of patients with complete response (CR) or partial response (PR) divided by all eligible and treated patients. Responses are evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) guideline. CR is defined as disappearance of all target and non-target lesions. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameters), and persistence of one or more non-target lesion(s).
Time Frame: as for outcome 1
Population: Eligible and treated patients.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm A (CE) | Arm B (CE+GDC-0449) | Arm C (CE+IMC-A12)
Number analyzed (Participants) | 48 | 52 | 52
Proportion of patients | 0.48 [0.33 to 0.63] | 0.56 [0.41 to 0.70] | 0.50 [0.36 to 0.64]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to death or date of last known alive.
Time Frame: Assessed every 3 months if patient is < 2 years from study entry, every 6 months if patient is 2-3 years from study entry
Population: Eligible and treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (CE) | Arm B (CE+GDC-0449) | Arm C (CE+IMC-A12)
Number analyzed (Participants) | 48 | 52 | 52
months | 8.8 [7.8 to 11.2] | 9.8 [8.7 to 12.4] | 10.1 [8.8 to 14.0]

4. Secondary Outcome: PFS
Description: Progression-free survival (PFS) is defined as the time from randomization to death or disease progression, whichever occurred first. Patients who were alive at the time of analysis are censored at the date at which they are last known to be alive and progression-free. This analysis is to evaluate the association between PFS and circulating tumor cells (CTCs).
Time Frame: as for outcome 1
Population: Eligible and treated patients who had baseline CTC results available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- High CTC Count: High CTC count is defined as greater than 100 CTCs per 7.5 ml at baseline.
- Low CTC Count: Low CTC count is defined as <= 100 CTCs per 7.5 ml at baseline.
Arm/Group | High CTC Count | Low CTC Count
Number analyzed (Participants) | 39 | 81
months | 4.1 [3.3 to 5.4] | 4.5 [4.4 to 5.3]
Statistical Analysis 1: Comparison: High CTC Count vs Low CTC Count; Test type: Superiority or Other; p = 0.01, Regression, Cox; Hazard Ratio (HR) = 1.69, 95% CI 2-sided [1.13 to 2.52] — Hazard ratio was derived comparing the high CTCs group to the low CTCs group

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment
Arm/Group | Arm A (CE) | Arm B (CE+GDC-0449) | Arm C (CE+IMC-A12)
Serious Adverse Events (participants affected / at risk) | 45/53 | 44/53 | 47/52
Other Adverse Events (participants affected / at risk) | 52/53 | 52/53 | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (CE) (N=53) | Arm B (CE+GDC-0449) (N=53) | Arm C (CE+IMC-A12) (N=52)
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 13 | 6 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 6 | 2
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Fatigue (General disorders) | 13 | 6 | 12
Fever (General disorders) | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 6
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 2
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 4
Nausea (Gastrointestinal disorders) | 6 | 6 | 11
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 3 | 7
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 0 | 1
Esophageal infection (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 2 | 3 | 1
Sepsis (Infections and infestations) | 0 | 1 | 2
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 2
Infections and infestations - Other (Infections and infestations) | 2 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Creatinine increased (Investigations) | 0 | 1 | 2
INR increased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 4 | 1 | 3
Neutrophil count decreased (Investigations) | 26 | 28 | 31
Platelet count decreased (Investigations) | 12 | 3 | 13
Weight loss (Investigations) | 0 | 3 | 3
White blood cell decreased (Investigations) | 25 | 23 | 27
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 2 | 6
Dehydration (Metabolism and nutrition disorders) | 7 | 2 | 7
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 5 | 1 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 7 | 7 | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal and connective - Other (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acoustic nerve disorder NOS (Nervous system disorders) | 0 | 0 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 3
Hypertension (Vascular disorders) | 0 | 2 | 0
Hypotension (Vascular disorders) | 3 | 0 | 1
Thromboembolic event (Vascular disorders) | 2 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (CE) (N=53) | Arm B (CE+GDC-0449) (N=53) | Arm C (CE+IMC-A12) (N=52)
Hearing impaired (Ear and labyrinth disorders) | 0 | 4 | 2
Tinnitus (Ear and labyrinth disorders) | 4 | 5 | 6
Anemia (Blood and lymphatic system disorders) | 39 | 43 | 46
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 0
Chills (General disorders) | 4 | 2 | 2
Edema limbs (General disorders) | 3 | 4 | 3
Fatigue (General disorders) | 38 | 46 | 42
Fever (General disorders) | 4 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 37 | 34 | 40
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1 | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 5 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 5 | 6
Abdominal pain (Gastrointestinal disorders) | 1 | 6 | 5
Constipation (Gastrointestinal disorders) | 18 | 20 | 18
Diarrhea (Gastrointestinal disorders) | 12 | 15 | 21
Dyspepsia (Gastrointestinal disorders) | 2 | 5 | 3
Mucositis oral (Gastrointestinal disorders) | 10 | 8 | 23
Nausea (Gastrointestinal disorders) | 33 | 31 | 35
Vomiting (Gastrointestinal disorders) | 19 | 16 | 19
Mucosal infection (Infections and infestations) | 0 | 3 | 2
Urinary tract infection (Infections and infestations) | 2 | 2 | 3
Alanine aminotransferase increased (Investigations) | 2 | 8 | 12
Alkaline phosphatase increased (Investigations) | 7 | 10 | 11
Aspartate aminotransferase increased (Investigations) | 1 | 5 | 11
Blood bilirubin increased (Investigations) | 1 | 1 | 3
Creatinine increased (Investigations) | 7 | 10 | 18
Lymphocyte count decreased (Investigations) | 5 | 6 | 5
Neutrophil count decreased (Investigations) | 12 | 14 | 11
Platelet count decreased (Investigations) | 28 | 23 | 34
Weight loss (Investigations) | 20 | 26 | 35
White blood cell decreased (Investigations) | 30 | 19 | 31
Investigations - Other, specify (Investigations) | 1 | 2 | 5
Anorexia (Metabolism and nutrition disorders) | 26 | 31 | 32
Dehydration (Metabolism and nutrition disorders) | 8 | 4 | 13
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 3 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 12 | 30
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 3 | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 11 | 16
Hypocalcemia (Metabolism and nutrition disorders) | 9 | 6 | 19
Hypokalemia (Metabolism and nutrition disorders) | 9 | 10 | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 19 | 21 | 21
Hyponatremia (Metabolism and nutrition disorders) | 17 | 14 | 17
Hypophosphatemia (Metabolism and nutrition disorders) | 7 | 5 | 4
Metabolism and nutrition - Other (Metabolism and nutrition disorders) | 2 | 2 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 6 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3
Musculoskeletal and connective - Other (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
Dizziness (Nervous system disorders) | 8 | 9 | 13
Dysgeusia (Nervous system disorders) | 10 | 18 | 13
Headache (Nervous system disorders) | 9 | 6 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 10 | 8
Blurred vision (Eye disorders) | 2 | 2 | 5
Insomnia (Psychiatric disorders) | 7 | 3 | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 4
Chronic kidney disease (Renal and urinary disorders) | 1 | 3 | 1
Hypertension (Vascular disorders) | 1 | 2 | 3
Hypotension (Vascular disorders) | 7 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less